CLINICAL TRIAL: NCT04252131
Title: Therapeutic Effect of Cassia Seed in Obesity of Patients With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Calo Psychiatric Center (Other)
Responsible Party: Principal Investigator, For-Wey Lung, superintendent, Calo Psychiatric Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 106-046
Record Dates: First submitted 2019-12-26; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Cassia seed; obesity; Therapeutic effect assessment; clinical trial
MeSH Terms: conditions — Schizophrenia; Obesity

STUDY DESIGN:
Intervention Model Description: Total of 92 schizophrenia patients with obesity was divided randomly into: 1) control group, received oral administration of Cassia seed placebo (3.0g), once/day for 12 weeks continuously; 2) treatment group, received oral administration of Cassia seed (3.0g), once/day for 12 weeks continuously.
Who Masked: Participant, Investigator
Masking Description: All participants are randomized into treatment or placebo group. Investigator also did not know who are in which group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cassia seed (Experimental): oral administration of Cassia seed (3.0g), once/day for 12 weeks
  Interventions: Drug: cassia seed tablet
- Cassia seed placebo (Placebo Comparator): oral administration of Cassia seed placebo (3.0g), once/day (90% of starch and 10% of cassia obtusifolia) for 12 weeks
  Interventions: Drug: cassia seed tablet

INTERVENTIONS:
Drug: cassia seed tablet — traditional Chinese herbs
  Other Names: cassia obtusifolia

SUMMARY:
Schizophrenia patients with anti-psychotics have decreased psychiatric symptoms, but have increased the generation of overweight or obesity. There is correlation between obesity, diabetes mellitus, metabolic syndrome, hypertension, hyperlipidemia and cardiovascular disorders. Cassia seed is one of traditional Chinese herbs, that can decline blood lipedema effect. Therefore, the purpose of the present study was to design a randomized, double blind, control group study to assess the therapeutic effect of Cassia seed in schizophrenia patients with obesity.

DETAILED DESCRIPTION:
Total of 92 schizophrenia patients with obesity will be enrolled and divided randomly into: 1) case group, received oral administration of Cassia seed (3.0g), once/day, 12 weeks; 2) control group, received oral administration of Cassia seed placebo (3.0g), once/day (90% of starch and 10% of cassia obtusifolia), 12 weeks. The primary outcome included the changes of body mass index (BMI), waist circumferences (WC); secondary outcome measured included the changes of hemoglobin A1c (HbA1c), total cholesterol, triglyceride, high density lipoprotein, low density lipoprotein, CRP (C-Reactive protein), IL-6, systolic blood pressure, diastolic blood pressure, and meridian energy.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 65 years
* diagnosed as schizophrenia at least more 6 months
* no major systemic illnesses based on physical examinations and laboratory test results
* BMI >= 24, WC >= 80 cm in female, WC >= 90 cm in male

Exclusion Criteria:

* participants were pregnant and lactating women
* allergy to Cassia
* SGOT or SGPT more than 2 times normal level
* BUN or creatinine more than normal level
* Fasting blood glucose (serum) > 140 mg/dL, systolic blood pressure > 180 mmHg, diastolic blood pressure > 110 mmHg, serum triglyceride > 400 mg/dL

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
physiological parameter for measuring Height and weight | 12 weeks
  the parameter of BMI in kg/m^2 for exploring the changes of body mass index (BMI) after cassia obtusifolia treatment
sphygmomanometer | 12 weeks
  the parameter of systolic blood pressure and diastolic blood pressure after cassia obtusifolia treatment

SECONDARY OUTCOMES:
Blood analyzer | 12 weeks
  the concentration of lipid profile, including total cholesterol, triglyceride, high denisty lipoprotein and low density lipoprotein after cassia obtusifolia treatment.
Meridian energy skin conductivity assessment using amperometer (0-200uA) | 12 weeks
  the parameter of meridian energy after cassia obtusifolia treatment

CONTACTS AND LOCATIONS:
Overall Officials: For-Wey Lung, MD, ScD, Principal Investigator — Calo Psychiatric Center
Locations (1):
- Calo Psychiatric Center, Pingtung City, Others, Taiwan